CLINICAL TRIAL: NCT06880640
Title: Affect-based Impulsivity in Borderline Personality Disorder: Developing a Neurocomputational Phenotype
Brief Title: Affect-based Impulsivity in Borderline Personality Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-3120; CTSC0406 (Other Grant/Funding Number: The North Carolina Translational and Clinical Sciences (TraCS) Institute)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Borderline Personality Disorder (BPD); Healthy Controls Group - Age and Sex-matched
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Psychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress (Experimental): Participants will undergo a controlled stress induction approximately 1 hour and 35 minutes into Session 1.
  Interventions: Behavioral: Stress Induction

INTERVENTIONS:
Behavioral: Stress Induction — Participants will complete the Trier Social Stress Test to induce stress, which includes a public speaking simulation and mental arithmetic.
  Other Names: Trier Social Stress Test (TSST)

SUMMARY:
The purpose of this research study is to investigate how personality traits and neuroendocrine systems relate to decision-making patterns in individuals 18-45 years old. The main question it aims to answer is how neuroendocrine activity impacts decision-making.

Participants will complete online behavioral tasks, a stress induction procedure, self-report surveys, and a cognitive assessment. During the session, psychophysiological measures will be collected, including electrocardiogram (ECG) and cardiac impedance (ICG) to monitor heart rate and blood flow, as well as electrodermal activity (EDA), blood drop samples, and saliva collection to assess nervous system activity.

ELIGIBILITY:
Inclusion Criteria:

Borderline Personality Disorder (BPD) group:

* Score of 38 or higher on Personality Assessment Inventory-Borderline Scale (PAI-BOR)
* Participants in the BPD group will be primarily recruited from the two

DEPENd lab studies that maintain large samples of BPD participants. To ensure maximal similarity between BPD participants recruited from other DEPENd lab studies and BPD participants recruited through other recruitment sources, the investigators will use the same criteria for the BPD group in the current study as the criteria used in the other DEPENd lab studies. BPD participants in the two DEPENd lab studies from which the investigators will be recruiting must meet the following criteria:

1. 3+ BPD symptoms, one of which must be affective instability, per clinical interview
2. Participants must score at least 80 on the Reynolds Intellectual Screening Test (RIST).

Health Control (HC) Group:

* Score of 12 or lower on PAI-BOR
* Score below 50th percentile on World Health Organization Disability Assessment Schedule (WHODAS)
* Absence of any current or lifetime psychiatric disorder, including personality disorders as determined by diagnostic interviews (SIDP and SCID), if the participant had participated in the lab's other studies (IRB Nos. 20-1735 and 21-0602).

Combined Inclusion Criteria:

* Ages 18-45
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Willingness to participate in all components of the study
* Participants must be able to speak, understand and read English.
* Participants must have at least 20/40 visual acuity (correct or uncorrected).

Exclusion Criteria:

* Use of as needed antihypertensive agents within 12 hours prior to lab visit
* Inability to refrain from using as needed psychotropic medications for 12 hours prior to lab visit
* History of psychotic disorder, Bipolar I disorder, autism spectrum disorder, reactive attachment disorder, pervasive developmental disorder, motor disorder, head injury, mental retardation, neurological disorder, or current substance dependence
* Family history of Bipolar I disorder in a first degree relative.
* Participants are also excluded for any of the following: cardiac pacemaker, aneurysm clip, cochlear implants, pregnancy, shrapnel, history of metal fragments in eyes, neurostimulators, weight of 250 lbs. or more, or claustrophobia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Goal-directed decision-making in the Social Decision Tree Task (SDTT) | Collected for 40 minutes ~2 hours into one-time study visit
  Measured by choice behavior in SDTT, which is based on the decision tree framework. After each action, participants receive feedback about the effect of that action and the extent to which it added to or took away from their points. If participants make a given choice, the subsequent actions that they can choose are different than if they were to initially make a different choice.
  An action in SDTT is goal-directed if the possible net gain an individual can earn before the end of the current epoch (a "day" in the SDTT) is equal to or higher than the amount they could gain by choosing the alternative action. The investigators will subset trials so that 1 is coded as choosing the immediately valuable action at the expense of the optimal and 0 is coded as choosing the optimal at the expense of the immediately valuable action. This outcome variable is binary.

SECONDARY OUTCOMES:
Bias toward social actions in the Social Decision Tree Task (SDTT) | Collected for 40 minutes ~2 hours into one-time study visit
  Measured by choice behavior in SDTT, which is based on the decision tree framework. An action in SDTT is defined as social if it is paired with a visual cue with a face on it and non-social if not. This outcome variable is binary.

OTHER OUTCOMES:
Change in salivary cortisol | Collected shortly after the participant consents into the study (~20 minutes into the one-time study visit) and 20 minutes after stress induction concludes (~2 hours into one-time study visit)
  The investigators will collect a saliva sample to measure baseline salivary cortisol at the beginning of the session. They will collect a second saliva sample 10 minutes after the stress induction concludes. They will measure cortisol levels in both samples through an assay. The investigators will calculate the change in salivary cortisol by subtracting the measured cortisol in the first saliva sample (collected at baseline) from the measured cortisol in the second saliva sample (collected 10 minutes after the stress induction). Salivary cortisol is measured as nmol/L. Salivary cortisol expected to generally be below 200 nmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallquist, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator who proposes to use the data has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Huys QJ, Eshel N, O'Nions E, Sheridan L, Dayan P, Roiser JP. Bonsai trees in your head: how the pavlovian system sculpts goal-directed choices by pruning decision trees. PLoS Comput Biol. 2012;8(3):e1002410. doi: 10.1371/journal.pcbi.1002410. Epub 2012 Mar 8. PMID 22412360